CLINICAL TRIAL: NCT05708638
Title: Does Anesthesia Induction With Target-controlled Infusion Reduce Post-induction Hypotension?
Brief Title: Target-controlled Infusion Anesthesia and Post-induction Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ATADEK 2022-18/04
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: General Anesthesia; Hemodynamic Instability
Keywords: General anesthesia; Target controlled infusion; Post-induction hypotension; Monitoring

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, non-blinded, randomized controlled trial, Patients were allocated to 2 groups:
  Group 1 Patients who underwent anesthesia induction with target-controlled infusion, Group 2: Patients who underwent manual anesthesia induction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who were assigned to have manual anesthesia induction group with propofol (Active Comparator): Patients who were assigned to have a manual anesthesia induction group, propofol was administered 2-3 mg/kg in 1-2 minutes to achieve a level of hypnosis measured by bispectral index ( BIS ) of 35-60.
  Interventions: Other: Manual anesthesia induction
- Patients who were assigned to have target controlled infusions ( TCI) induction with propofol (Active Comparator): Patients who were assigned to have TCI induction had the target effect site concentration (Ce) of propofol (Ce) set at 3 μg ml-1 using the Schneider model and subsequently modified to achieve and maintain a level of hypnosis measured by BIS of 35-55
  Interventions: Other: Anesthesia induction with Target controlled infusions (TCI)

INTERVENTIONS:
Other: Manual anesthesia induction — In manual anesthesia induction, anesthetic agents are administered at a fixed dose and rate adjusted according to the patient's weight
  Other Names: Manuel induction
  Arms: Patients who were assigned to have manual anesthesia induction group with propofol
Other: Anesthesia induction with Target controlled infusions (TCI) — Target controlled infusion (TCI) system aims to reach the theoretically targeted blood or brain concentration of anesthetic agents based on the patient's age, weight, and height, with computer-assisted algorithms.
  Other Names: TCI induction
  Arms: Patients who were assigned to have target controlled infusions ( TCI) induction with propofol

SUMMARY:
Hemodynamic changes during induction of anesthesia may have adverse outcomes and should therefore be avoided. The decrease in blood pressure during induction of anesthesia with propofol is due to a decrease in systemic vascular resistance or cardiac output and may be increased by the concomitant use of other drugs such as remifentanil. Target controlled infusion (TCI) system aims to reach the theoretically targeted blood or brain concentration of anesthetic agents based on the patient's age, weight, and height, with computer-assisted algorithms. In manual anesthesia induction, anesthetic agents are administered at a fixed dose and rate adjusted according to the patient's weight, which may cause hypotension in patients with low cardiovascular performance. As target-controlled infusion (TCI) obviates the need to calculate the infusion rate manually, the use of TCI may provide a better hemodynamic profile during anesthesia induction This study was designed to test the hypothesis that propofol by TCI anesthesia induction is associated with a lower hypotension rate when compared with manual anesthesia induction

DETAILED DESCRIPTION:
Maintaining normotension is one of the top priorities for anesthesiologists due to its negative effects. Although there are a lot of studies and knowledge on the topic approximately 20-30% of patients develop post-induction hypotension. Mostly it occurs due to the adverse effects of anesthetics such as a decrease in systemic vascular resistance or cardiac output and the interplay between them. The risk can be minimized in two steps: first by identifying high-risk patients, and second with tight control of hemodynamic parameters. As a second step, tight hemodynamic control during induction may be done using target-controlled infusion (TCI) systems, which systems help to adjust the dosage to the needs of each patient by measuring hypnotic effects through the bispectral index (BIS).

TCI models for propofol have been previously compared with manual infusions, however, it is not clear whether it still contributes to or triggers hemodynamic deterioration. Therefore in this study, the investigators' aim is to determine the effect of two different anesthesia techniques on the development of postinduction hypotension through hemodynamic parameters monitored by the pressure recording analytical method (PRAM). The secondary aim is to identify risk factors that can predict postinduction hypotension

ELIGIBILITY:
Inclusion Criteria:

* Patients with the American Society of Anesthesiology physical status 1-3
* Underwent major elective surgery
* Required intra-arterial blood pressure monitoring before induction.

Exclusion Criteria:

* Under 18 years of age
* Arrhythmia (atrial fibrillation, frequent premature beat)
* Severe valvular heart disease
* Morbid obesity
* Intubation difficulty
* Drug addiction
* Treatment with opiates
* Pregnancy
* Emergency surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Systolic arterial pressure (SAP), measured before and after anesthesia induction was assessed to determine of post-induction hypotension in patients undergoing general anesthesia induction with TCI (target controlled infusion) or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Systolic arterial pressure (SAP- mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SAP is a parameter used to assess the pressure of the arterial system during cardiac systole
Diastolic arterial pressure (DAP), measured before and after anesthesia induction was assessed to determine of post-induction hypotension in patients undergoing general anesthesia induction with TCI (target controlled infusion) or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Diastolic arterial pressure (DAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). DAP is a parameter used to assess the pressure of the arterial system during cardiac diastole.
Mean arterial pressure (MAP), measured before and after anesthesia induction was assessed to determine of post-induction hypotension in patients undergoing general anesthesia induction with TCI (target controlled infusion) or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Mean arterial pressure (MAP, mm/Hg) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). MAP is a parameter used to assess organ perfusion

SECONDARY OUTCOMES:
Arterial elastance (Ea) measured before anesthesia induction was investigated whether is a predictive parameter for post-induction hypotension in patients undergoing general anesthesia with TCI or manual | he duration of the study was defined from one minute before induction to 10 minutes after induction
  Ea ((mmHg m-2ml-1)is an indicator of cardiac afterload and arterial tone and can be calculated by the ratio of the end-systolic pressure (ESP) and stroke volume (SV) obtained from arterial wave analysis. Ea was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy) before the anesthesia induction
Stroke volume variation (SVV), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI and manual | The duration of the study was defined from one minute before induction to 10 minutes after induction]
  Stroke volume variation (SVV,%), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). SVV is a parameter used to asses cardiac preload and fluid responsiveness
Pulse pressure variation (PPV), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Pulse pressure variation (PPV,%) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). PPV is a parameter used to asses cardiac preload and fluid responsiveness.
Cardiac power output (CPO), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Cardiac power output (CPO, Watt) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CPO is a parameter used to asses cardiac reserve
Cardiac index (CI), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Cardiac index (CI, L/min/m2), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). CI is a parameter used to asses cardiac stroke volume
Dp/Dt, measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Dp/Dt(mmHg/msn), was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). Dp/Dt is a parameter used to asses cardiac contractility.
Heart rate (HR), measured before anesthesia induction were assessed for prediction of post-induction hypotension in patients undergoing general anesthesia induction with TCI or manual | The duration of the study was defined from one minute before induction to 10 minutes after induction
  Heart rate (HR/bpm) was monitored using the uncalibrated pulse contour device MostCare (Vytech, Vygon, Padova, Italy). HR is a parameter used to assess the cardiac rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Mu J, Jiang T, Xu XB, Yuen VM, Irwin MG. Comparison of target-controlled infusion and manual infusion for propofol anaesthesia in children. Br J Anaesth. 2018 May;120(5):1049-1055. doi: 10.1016/j.bja.2017.11.102. Epub 2018 Feb 3. PMID 29661382
- [Background] Hsieh ML, Lu YT, Lin CC, Lee CP. Comparison of the target-controlled infusion and the manual infusion of propofol anesthesia during electroconvulsive therapy: an open-label randomized controlled trial. BMC Psychiatry. 2021 Feb 4;21(1):71. doi: 10.1186/s12888-021-03069-6. PMID 33541306
- [Result] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Result] Guarracino F, Lapolla F, Cariello C, Danella A, Doroni L, Baldassarri R, Boldrini A, Volpe ML. Target controlled infusion: TCI. Minerva Anestesiol. 2005 Jun;71(6):335-7. PMID 15886597
- [Result] Leslie K, Clavisi O, Hargrove J. Target-controlled infusion versus manually-controlled infusion of propofol for general anaesthesia or sedation in adults. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD006059. doi: 10.1002/14651858.CD006059.pub2. PMID 18646134
- [Result] Marik PE. Noninvasive cardiac output monitors: a state-of the-art review. J Cardiothorac Vasc Anesth. 2013 Feb;27(1):121-34. doi: 10.1053/j.jvca.2012.03.022. Epub 2012 May 19. No abstract available. PMID 22609340